CLINICAL TRIAL: NCT06773091
Title: An Open-Label, Single-Arm, Multicenter Phase I Clinical Study to Evaluate the Safety and Preliminary Efficacy of NK042 Cell Injection (Universal NKR+NK) in Advanced Solid Tumors
Brief Title: A Phase I Study of NK042 Cell Injection in Advanced Solid Tumors
Acronym: NKSOLID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai NK Cell Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK042-I-ST-01
Record Dates: First submitted 2025-01-06; First posted 2025-01-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors
Keywords: CAR-NK; Advanced solid tumors; Early-phase clinical trial; Cell Therapy
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK042 - cellular therapy (Experimental): Phase Ia (Dose Escalation): Determines maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) using single- and multiple-dose escalation with a "3+3" design.
  Phase Ib (Cohort Expansion): Evaluates safety, tolerability, and efficacy in solid tumor indications that demonstrated preliminary efficacy in Phase Ia.
  Participants undergo lymphodepletion prior to the first infusion of NK042.
  Interventions: Biological: NK042; Drug: Fludarabine (FLU); Drug: Cyclophosphamide (CTX)

INTERVENTIONS:
Biological: NK042 — NK042 is an allogeneic, off-the-shelf cellular therapy derived from healthy donors and enriched with NKR+ NK cells.
Drug: Fludarabine (FLU) — Fludarabine (FLU) is administered as a lymphodepletion regimen prior to NK042 infusion.
Drug: Cyclophosphamide (CTX) — Cyclophosphamide (CTX) is administered as a lymphodepletion regimen prior to NK042 infusion.

SUMMARY:
This is a single-arm, open-label, multi-center phase 1 clinical study designed to evaluate the safety and preliminary efficacy of NK042 cell injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is divided into two phases: Phase Ia and Phase Ib.

Dose-Escalation and Expansion:

* Phase Ia: This dose-escalation phase involves both single-dose and multiple-dose administrations of NK042 in patients with advanced solid tumors.
* Phase Ib: This multiple-dose cohort-expansion phase will focus on solid tumor indications that demonstrated preliminary efficacy in Phase Ia.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of a written informed consent form.
2. Age between 18 and 70 years.
3. Histologically or cytologically confirmed locally advanced or metastatic solid tumor patients who are not amenable to surgical resection, with no standard treatment options, or who have relapsed or progressed after standard treatment, or are resistant or intolerant to standard treatment.
4. At least one assessable tumor lesion according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Expected survival ≥12 weeks.
7. Must have adequate bone marrow, liver, and renal function.

Exclusion Criteria:

1. Insufficient washout period for prior anti-tumor treatments before the first dose, including chemotherapy, targeted therapy, antibody therapy, and radiotherapy.
2. Participation in another clinical trial and use of investigational drugs within 28 days before the first dose.
3. Requirement for anticoagulation therapy.
4. Symptomatic brain parenchymal metastases with less than 4 weeks of stability after treatment.
5. Active pulmonary diseases, including but not limited to interstitial lung disease, pneumonitis.
6. Uncontrolled active infections.
7. Uncontrollable massive pleural effusion, ascites, or pericardial effusion.
8. Previous receipt of other cellular therapies.
9. Planned concurrent participation in other anti-tumor treatments during the study.
10. Pregnant or breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events (AEs) and Serious Adverse Events (SAEs) | Up to 1 year after first dose of NK042.
  Number of subjects experiencing adverse events, and the frequency and severity of adverse events. The type, frequency, onset, and severity of treatment-emergent adverse events (TEAEs) will be assessed in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE),version 5.0.
Dose Limiting Toxicities (DLTs) | Up to 28-day after first dose of NK042.
  Identification of DLTs to determine the maximum tolerated dose (MTD).
Objective Response Rate (ORR) | Up to 1 year after first dose of NK042.
  The proportion of participants achieving a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Predose, 4, 24, 48, 72, Day 8, Day 15, Day 22, Day 29 post-dose and every 2 months during the treatment follow-up period.
  Cmax of NK042 will be measured to determine the maximum concentration reached in the plasma following administration.
Time to reach maximum concentration (Tmax) | Predose, 4, 24, 48, 72 hours, Day 8, Day 15, Day 22, Day 29 post-dose, and every 2 months during the treatment follow-up period.
  Tmax of NK042 will be assessed to determine the time point at which the highest plasma concentration is observed following administration.
Area under the plasma concentration versus time curve (AUC₀-ₜ) | Predose, 4, 24, 48, 72 hours, Day 8, Day 15, Day 22, Day 29 post-dose, and every 2 months during the treatment follow-up period.
  AUC₀-ₜ will be assessed to determine the total NK042 exposure from the time of administration (0) to the last measurable concentration (t).
Half-life (T₁/₂) of NK042 | Predose, 4, 24, 48, 72 hours, Day 8, Day 15, Day 22, Day 29 post-dose, and every 2 months during the treatment follow-up period.
  T₁/₂ of NK042 will be assessed to determine the time required for a 50% reduction in the maximum amount of circulating NK042 in the plasma.
Progression-Free Survival (PFS) | Up to 1 year after first dose of NK042 .
  The time from the first dose until objective tumor progression or death.
Overall Survival (OS) | Up to 1 year after first dose of NK042 .
  The time from the first dose until death from any cause.
Duration of Response (DOR) | Up to 1 year after first dose of NK042 .
  The time from the first documentation of CR or PR to disease progression or death.
Disease Control Rate (DCR) | Up to 1 year after first dose of NK042 .
  The proportion of participants who achieve a CR, PR, or stable disease (SD) as assessed by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No